CLINICAL TRIAL: NCT04836078
Title: Performance of Simvastatin Microsponges as a Local Treatment for Chronic Periodontitis - Randomized Clinical Trial
Brief Title: Role of Simvastatin Microsponges in Treatment of Periodontitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mortada, Lecturer at the Department of Periodontology and Oral Implantology , Faculty of Dentistry , Assiut University, Egypt, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Simvastatin in periodontitis
Record Dates: First submitted 2021-03-25; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Gels

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plain chitosan gel group (Placebo Comparator): After the reevaluation phase after that corrective surgical phase started for the three groups. Local infiltration anesthesia administrated then sulcular flaps raised for the purpose of open flap subgingival debridement . Randomization will be performed and concealment from the assessors. For root conditioning purpose, Group (I) ; will be injected subgingivally with chitosan 2% gel .
  Interventions: Procedure: open flap subgingival debridement; Procedure: Subgingival injection of chitosan 2% gel
- Chitosan gels containing free Simvastatin (Active Comparator): Will be injected subgingivally with simvastatin microsponges dispersed into chitosan 2% gel. .
  Interventions: Procedure: open flap subgingival debridement; Procedure: Subgingival injection of chitosan 2% gel
- Chitosan gels containing Simvastatin microsponges (Experimental): This group will be injected subgingivally with free simvastatin dispersed into chitosan 2% gel containing .
  Interventions: Procedure: open flap subgingival debridement; Procedure: Subgingival injection of chitosan 2% gel

INTERVENTIONS:
Procedure: open flap subgingival debridement — After the reevaluation phase after that corrective surgical phase started for the three groups. Local infiltration anesthesia administrated then sulcular flaps raised for the purpose of open flap subgingival debridement.Randomization was then performed and concealment from the assessors.
Procedure: Subgingival injection of chitosan 2% gel — Group (I); injected subgingivally with chitosan 2% gel containing a microsponges formulated drug weekly
  Arms: Plain chitosan gel group
Procedure: Subgingival injection of chitosan 2% gel — Group (II); injected subgingivally with chitosan 2% gel containing free drug weekly
  Arms: Chitosan gels containing free Simvastatin
Procedure: Subgingival injection of chitosan 2% gel — Group (III); injected subgingivally with placebo chitosan 2% gel weekly
  Arms: Chitosan gels containing Simvastatin microsponges

SUMMARY:
the aim of our study is to enhance the dissolution and subsequently the local penetration of the drug through the sulcus in addition to controlling the drug release so that, the drug could be potentially absorbed.

DETAILED DESCRIPTION:
Patients will be divided randomly into three groups: Group (I);will be treated with subgingival debridement and subgengival injection of chitosan 2% gel containing a microsponges formulated (SV), Group (II); will be treated with subgingival debridement and subgingival injection of chitosan 2% gel containing free (SV) and Group (III); will be treated by subgingival debridement and placebo gel injected subgingivally. Pocket depth and clinical attachment loss bone gain were recorded preoperative and six months postoperative for all groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic periodontitis with minimum two sites of pocket depth > 5 mm
* patients with normal lipid profile
* nonsmokers
* patients free from any systemic disorders
* committed patients to complete the treatment with follow-ups.

Exclusion Criteria:

* patients with hyperlipidemia
* patients taking lipid lowering drugs
* smokers
* pregnant
* Lactating women women, patients with mental or psychological illness and medically compromised patients.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Pocket depth | Before the beginning of study
  Will be measured in millimetre
Pocket depth | By the end of study after 6 months of 6 months
  Will be measured in millimetre
Clinical attachment loss | Before beginning of the study
  Will be measured in millimetre
Clinical attachment loss | By the end of study after 6 months of 6 months
  Will be measured in millimetre

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No